CLINICAL TRIAL: NCT07265050
Title: Comparison of Emergence Agitation Between Remimazolam With Flumazenil and Propofol-based Total Intravenous Anesthesia in Patients Undergoing Nasal Surgery: A Randomized Controlled Trial
Brief Title: Comparison of Emergence Agitation Between Remimazolam With Flumazenil and Propofol-based Total Intravenous Anesthesia in Patients Undergoing Nasal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2507-174-1661
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — remimazolam; Flumazenil; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): Participants receive general anesthesia induced and maintained with remimazolam-based total intravenous anesthesia. At the end of surgery, flumazenil (0.2-1.0 mg) is administered to reverse the sedative effect.
  Interventions: Drug: Remimazolam with Flumazenil
- Propofol (Active Comparator): Participants receive general anesthesia induced and maintained with propofol.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam with Flumazenil — General anesthesia is induced and maintained with remimazolam (initial infusion approximately 6 mg/kg/hr for induction, then 1-2 mg/kg/hr for maintenance), along with remifentanil for analgesia. At the end of surgery, flumazenil is administered to reverse the sedative effect, starting with 0.2 mg IV, followed by 0.1 mg incremental doses every 1 minute as needed, up to a total dose of 1.0 mg.
  Arms: Remimazolam
Drug: Propofol — General anesthesia is induced and maintained with propofol using target-controlled infusion (effect-site concentration up to 4.0 μg/mL), along with remifentanil for analgesia.
  Arms: Propofol

SUMMARY:
Participants will be randomly assigned to receive general anesthesia with either remimazolaml-based total intravenous anesthesia reversed with flumazenil or propofol-based total intravenous anesthesia. The primary outcome is the incidence of emergence agitation evaluated at the time of awakening after surgery. Additional outcomes include time to extubation, hemodynamic stability, airway complications such as coughing or laryngospasm, and postoperative recovery profiles including pain, nausea, vomiting, and sedation in the post-anesthesia care unit. This study aims to determine whether remimazolam with flumazenil provides smoother emergence compared with propofol in patients undergoing nasal surgery.

ELIGIBILITY:
Inclusion Criteria

- Adults aged 19 years or older scheduled to undergo nasal surgery requiring general anesthesia

Exclusion Criteria

* Declines or is unable to provide informed consent
* Body mass index (BMI) ≥ 30 kg/m²
* Pre-existing neurological or cognitive impairment
* Known contraindication or allergy to remimazolam, propofol, or flumazenil
* Any condition judged by the investigator to make participation inappropriate (e.g., unstable medical status, severe comorbidities)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Emergence Agitation | From discontinuation of anesthesia to exit in the operating room

SECONDARY OUTCOMES:
Time to Tracheal Extubation | From anesthesia discontinuation to extubation in the operating room
Intraoperative Hemodynamic Stability | During anesthesia
Incidence of Airway Complications During Emergence | during anesthesia
  Complications such as coughing, desaturation, and laryngospasm will be recorded based on direct observation by anesthesiologists.